CLINICAL TRIAL: NCT01046708
Title: Ovulation Induction With Clomiphene Citrate: to Support or Not to Support the Luteal Phase
Brief Title: Luteal Support and Intrauterine Insemination (IUI) With Clomiphene Citrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Kyrou Dimitra, Doctor, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFER
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Infertility
Keywords: IUI; clomiphene citrate; utrogestan
MeSH Terms: conditions — Infertility | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- micronized progesterone (Experimental)
  Interventions: Drug: micronized progesterone
- no utrogestan (No Intervention)

INTERVENTIONS:
Drug: micronized progesterone — 600mg in 3 separate doses per day
  Other Names: utrogestan
  Arms: micronized progesterone

SUMMARY:
The purpose of this study is to assess the effect of luteal phase supplement (LPS) on pregnancy rate in IUI cycles stimulated with clomiphene citrate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 36 years
* Body mass index between 18 and 29
* Presence of both ovaries
* Basal levels of estradiol (≤ 80 pg/ml) and progesterone (≤ 1.6ng/ml) on day one of the cycle and a day three FSH level of <12IU/L
* Patients can enter the study only once.
* Only the first IUI attempt will be included ( at the 2nd and 3 rd attempt progesterone could be administrated if it is necessary but these attempts will be excluded from the study)
* Normal HSG (maximum 3 months prior starting the stimulation).
* Donor sperm can be included

Exclusion Criteria:

* Polycystic ovarian syndrome (Rotterdam criteria)
* Endometriosis(≥AFS III)

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 1 year

SECONDARY OUTCOMES:
implantation rate,clinical pregnancy rate | 1 year

REFERENCES:
- [Derived] Kyrou D, Fatemi HM, Tournaye H, Devroey P. Luteal phase support in normo-ovulatory women stimulated with clomiphene citrate for intrauterine insemination: need or habit? Hum Reprod. 2010 Oct;25(10):2501-6. doi: 10.1093/humrep/deq223. Epub 2010 Aug 18. PMID 20719809